CLINICAL TRIAL: NCT05030519
Title: A Study of Diarrhea and Intestinal Flora Changes Caused by Pyrotinib in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: intestinal flora study
Record Dates: First submitted 2021-08-25; First posted 2021-09-01 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Trastuzumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Identify the abundance of intestinal flora and the number of bacteria through metagenomic sequencing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib 400 mg once daily(monotherapy or combined Trastuzumab/Inetetamab and chemotherapy)
  Other Names: Trastuzumab/Inetetamab and other chemotherapy

SUMMARY:
By measuring the intestinal flora abundance and bacterial count of patients in the early stage of using pyrotinib to clarify the relationship between diarrhea caused by pyrotinib and changes in intestinal flora in breast cancer patients, the correlation between the change of intestinal flora and the relief of diarrhea are also explored after two-cycle treatment.

DETAILED DESCRIPTION:
In recent years, small-molecule tyrosine kinase inhibitors (TKI) have achieved good results in anti-HER2 therapy and have been widely used in clinical practice, such as Breast cancer. However, such drugs can easily cause diarrhea and disorders of intestinal flora , may affect the efficacy of the drug and lead to the occurrence of other diseases.This study is to clarify the connection between the diarrhea caused by pyrotinib and the change of intestinal flora, pave the way for studying on whether the flora affects the efficacy of the drug and whether the flora should be supplemented appropriately in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Female breast cancer patients aged 18-75 years.
2. ECOG performance status of 0 to 1;
3. Known hormone receptor status;
4. HER2 positive breast cancer and previously reveived ≤2 anti-HER2 therapy;
5. Breast cancer patients are about to receive pyrotinib monotherapy or combined with Trastuzumab/Inetetamab and chemotherapy；
6. Patients with adequate organ function before enrollment (no blood transfusion, no white blood cell or platelet-elevating drugs used within 2 weeks before screening): 1) Blood routine:ANC≥1.5×10^9/L; PLT≥90×10^9/L; Hb≥90 g/L；2)Blood biochemistry: TBIL≤1.5×ULN;ALT and AST ≤1.5×ULN; alkaline phosphatase ≤ 2.5×ULN; BUN and Cr≤1.5×ULN；3) Cardiac color Doppler ultrasound:LVEF≥55%；4) 12-lead ECG: QTcF < 470 msec;
7. Signed the informed consent form prior to patient entry, and have good compliance and are willing to cooperate with follow-up.

Exclusion Criteria:

1. patients with Severe heart disease or discomfor;
2. Previous or ongoing use of HER2-targeted tyrosine kinase inhibitors ;
3. Inability to swallow, intestinal obstruction, or other factors that affect the taking and absorption of the drug;
4. Allergy to pyrotinib; history of immunodeficiency, including HIV positive, active HBV/HCV, other acquired or congenital immunodeficiency disease and organ transplantation history;
5. Patients during pregnancy or lactation, patients with childbearing potential tested positive in baseline pregnancy test, or patients unwilling to take effective contraceptive measures throughout the trial and 7 months after the last study medication;
6. patients with intestinal disease, serious concomitant diseases, or other comorbid diseases that will interfere with the planned treatment, or patients not eligible for this study judged by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2-positive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The quantity of intestinal flora from breast cancer patients' fecal microflora at different follow-up nodes | January 2021- December 2022
  Fecal samples were collected from patients at each follow-up node to detect the number of bacterial species in the intestinal flora
The abundance of intestinal flora from breast cancer patients' fecal microflora at different follow-up nodes | January 2021- December 2022
  Fecal samples were collected at each follow-up node to detect the richness of different bacterial species in intestinal flora

SECONDARY OUTCOMES:
Disease Control Rate（DCR） | January 2021- December 2022
  DCR=CR+PR+SD Complete Remission(CR): All target lesions disappeared, no new lesions appeared, and tumor markers were normal, for at least 4 weeks; Partial Remission(PR): The sum of the maximum diameter of the target lesion is reduced by ≥30% and maintained for at least 4 weeks; Stable Disease(SD): The maximum diameter and reduction of the target lesion did not reach the PR, or the enlargement did not reach the PD;
Overall Survival（OS） | January 2021- December 2022
  Time interval from randomization to death for any reason
Progression Free Survival (PFS) | January 2021- December 2022
  Time interval from randomization to first disease progression or death for any reason
Objective Response Rate (ORR) | January 2021- December 2022
  ORR=CR+PR Complete Remission(CR): All target lesions disappeared, no new lesions appeared, and tumor markers were normal, for at least 4 weeks; Partial Remission(PR): The sum of the maximum diameter of the target lesion is reduced by ≥30% and maintained for at least 4 weeks;

CONTACTS AND LOCATIONS:
Overall Officials: Wenming Cao, Ph.D., Principal Investigator — Department of Breast Medical Oncology, Zhejiang Cancer Hospital
Locations (1):
- China, Zhejiang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ross JS. Breast cancer biomarkers and HER2 testing after 10 years of anti-HER2 therapy. Drug News Perspect. 2009 Mar;22(2):93-106. doi: 10.1358/dnp.2009.22.2.1334452. PMID 19330168
- [Result] Freudenberg JA, Wang Q, Katsumata M, Drebin J, Nagatomo I, Greene MI. The role of HER2 in early breast cancer metastasis and the origins of resistance to HER2-targeted therapies. Exp Mol Pathol. 2009 Aug;87(1):1-11. doi: 10.1016/j.yexmp.2009.05.001. Epub 2009 May 18. PMID 19450579
- [Result] Ley RE, Peterson DA, Gordon JI. Ecological and evolutionary forces shaping microbial diversity in the human intestine. Cell. 2006 Feb 24;124(4):837-48. doi: 10.1016/j.cell.2006.02.017. PMID 16497592
- [Result] Fernandez MF, Reina-Perez I, Astorga JM, Rodriguez-Carrillo A, Plaza-Diaz J, Fontana L. Breast Cancer and Its Relationship with the Microbiota. Int J Environ Res Public Health. 2018 Aug 14;15(8):1747. doi: 10.3390/ijerph15081747. PMID 30110974
- [Result] Parida S, Sharma D. The power of small changes: Comprehensive analyses of microbial dysbiosis in breast cancer. Biochim Biophys Acta Rev Cancer. 2019 Apr;1871(2):392-405. doi: 10.1016/j.bbcan.2019.04.001. Epub 2019 Apr 11. PMID 30981803
- [Result] Yang J, Tan Q, Fu Q, Zhou Y, Hu Y, Tang S, Zhou Y, Zhang J, Qiu J, Lv Q. Gastrointestinal microbiome and breast cancer: correlations, mechanisms and potential clinical implications. Breast Cancer. 2017 Mar;24(2):220-228. doi: 10.1007/s12282-016-0734-z. Epub 2016 Oct 5. PMID 27709424
- [Result] Ma H, Bernstein L, Pike MC, Ursin G. Reproductive factors and breast cancer risk according to joint estrogen and progesterone receptor status: a meta-analysis of epidemiological studies. Breast Cancer Res. 2006;8(4):R43. doi: 10.1186/bcr1525. PMID 16859501
- [Result] Gaudet MM, Gierach GL, Carter BD, Luo J, Milne RL, Weiderpass E, Giles GG, Tamimi RM, Eliassen AH, Rosner B, Wolk A, Adami HO, Margolis KL, Gapstur SM, Garcia-Closas M, Brinton LA. Pooled Analysis of Nine Cohorts Reveals Breast Cancer Risk Factors by Tumor Molecular Subtype. Cancer Res. 2018 Oct 15;78(20):6011-6021. doi: 10.1158/0008-5472.CAN-18-0502. Epub 2018 Sep 5. PMID 30185547
- [Result] Wu AH, Tseng C, Vigen C, Yu Y, Cozen W, Garcia AA, Spicer D. Gut microbiome associations with breast cancer risk factors and tumor characteristics: a pilot study. Breast Cancer Res Treat. 2020 Jul;182(2):451-463. doi: 10.1007/s10549-020-05702-6. Epub 2020 May 28. PMID 32468338
- [Result] Goedert JJ, Jones G, Hua X, Xu X, Yu G, Flores R, Falk RT, Gail MH, Shi J, Ravel J, Feigelson HS. Investigation of the association between the fecal microbiota and breast cancer in postmenopausal women: a population-based case-control pilot study. J Natl Cancer Inst. 2015 Jun 1;107(8):djv147. doi: 10.1093/jnci/djv147. Print 2015 Aug. PMID 26032724